CLINICAL TRIAL: NCT03336749
Title: SENSory Re-learning of the UPPer Limb After Stroke (SENSUPP): a Pilot Randomized Controlled Trial
Brief Title: Sensory Re-learning of the Upper Limb After Stroke
Acronym: SENSUPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Christina Brogardh, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sensory
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: Stroke, upper limb, sensory training, rehabilitation
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: The assessors are blinded to the participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory group (Experimental): Sensory re-learning in combination with task-specific training
  Interventions: Behavioral: Sensory group
- Control group (Active Comparator): Traditional task-specific training
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Sensory group — The sensory re-learning consists of touch detection practice, i.e., touch discrimination to identify different materials, shapes, textures, weights and temperatures, proprioception and tactile object recognition in combination with task-specific training.
  Arms: Sensory group
Other: Control group — Traditional task-specific training
  Arms: Control group

SUMMARY:
The overall aim of this study is to investigate if sensory re-learning in combination with task-specific training is more effective than task-specific training alone to improve sensory function of the hand, dexterity, the ability to use the hand in daily activities, perceived participation and life satisfaction.

DETAILED DESCRIPTION:
More than half of stroke survivors suffer from sensory impairments of their affected upper limb (UL), which can lead to long term problems to use the UL in daily life, such as personal care, household- and leisure activities. Few studies have evaluated if sensory re-learning in combination with task-specific training can improve the ability to perform daily hand activities and perceived participation. Therefore, there is a need for more studies. This is a single-blinded pilot randomized controlled trial with two treatment arms. Thirty persons with sensory impairments of the UL after stroke will be recruited and randomized to either sensory re-learning in combination with task-specific training or to task-specific training only. The training will consist of 2.5 hours of group training per session, 2 times per week for 5 weeks. Assessments will be conducted pre- and post-training and at 3 months' after the intervention.

Descriptive statistics (mean (SD) or median (min- max) will be used to characterize the study groups. Non-parametric statistics will be used for ordinal data and parametric statistics for continues data. To analyze between group differences, the Mann-Whitney test or Independent sample t-test will be used and Wilcoxon signed ranks test or paired t-test to analyze within group differences. The level of statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* sensory impairments (≤5 points in Shape-Texture Identification test) of upper limb after stroke
* ability to grasp and release an object
* be able to understand oral and written information
* 18-80 years of age
* at least 6 months since stroke onset
* be able to walk with or without an assistive device

Exclusion Criteria:

• sensory impairments of the UL due to other diagnosis than stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Change in Semmes- Weinstein monofilament (SWM) test from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 months.
  Assess touch detection thresholds of the hand and fingers. The short version with 5 filaments from 0.07 gram to 279 grams will be used. The touch detection thresholds are scored on a 0 to 5-point scale, where 5 represents the thinnest filament and 0 represents the largest filament. Five different positions of the hand are tested: fingertip on digit I, II, V and on the thenar and hypothenar region. Both hands are tested and the total sum score is 25 for each hand.
Change in Shape- Texture Identification test (STI) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 months.
  Measures the ability to identify shapes and textures. Both the affected and non- affected hand are tested and the scores range from 0 to 3 points per hand for each subtest with a maximum score of 6 points.
Change in Fugl- Meyer Assessment (FMA-UE) sensory section from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 months.
  Measures light touch and proprioception of the upper limb after stroke. The score ranges from 0 to 4 points for each subtest with a maximum score of 8 points per hand.
Change in Tactile object identification test from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 months.
  Measures the ability to identify different objects without vision. Out of 20 objects, 15 are used during the assessment. Within 15 seconds the participant should blind-fold recognize an object. Correct answer yields 2 points, recognition of some feature of the object yields 1 point and incorrect answer 0 points; thus a maximum total sum score of 30 points.

SECONDARY OUTCOMES:
Change in Box and Block Test (BBT) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Measures gross manual dexterity. It consists of a box with two compartments and of 100 wooden blocks. The number of blocks that can be transported from one compartment to the other during 1 minute is counted.
Change in Mini Sollerman Hand Function Test (mSHFT) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Measures fine motor dexterity. It consists of three tasks: (1) picking up four coins from a purse, (2) putting four nuts on bolts and (3) buttoning four buttons in decreasing sizes. The score ranges from 0 to 4 points for each task with a maximum score of 12 points.
Change in Modified Motor Assessment Scale (M-MAS) for the upper limb from baseline to post intervention and from baseline to 3 month follow-up.. | Baseline, 5 weeks, 3 month.
  Measures fine motor dexterity. The scale ranges from 0 to 5 points where 0 point represents no motor function and 5 points represents almost normal or normal motor function.
Change in Grippit from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Grip strength, the highest isometric contraction of three trials is recorded in Newton (N).
Changes in Motor Activity Log (MAL) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Measures activity in daily living with a 30-item scale where the participants rate how much (amount of use; AOU) and how well (quality of movement; QOM) they use their affected hand in daily activities. The score ranges from 0 (never use the affected arm for this activity) to 5 (always use the affected arm for this activity) and for QOM from 0 (inability to use the affected arm for this activity) to 5 (ability to use the affected arm for this activity just as well as before the stroke).
Change in Canadian Occupational Performance Measure (COPM) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Perceived difficulties in daily activities. This is a client-centered interview based outcome measure, where the participants identify problems in their execution of activities in self-care, productivity and leisure activities. The self-perceived performance and satisfaction of their sensory related problems are rated on a scale ranging from 1 (not able to do respective not satisfied) to 10 (able to do extremely well respective extremely satisfied). Higher ratings indicate better performance and more satisfaction.
change in Stroke Impact Scale, (SIS) Participation domain from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  It measures a person's perceived participation through eight items, i.e., how stroke impact on work, social activities, quiet recreations, active recreations, role as a family member, religious activities, life control and ability to help others. Every item is scored on a 5- grade scale from 5 (none of the time) to 1 (all of the time).
Change in Life Satisfaction Scale (LiSat) from baseline to post intervention and from baseline to 3 month follow-up. | Baseline, 5 weeks, 3 month.
  Measures life satisfaction. In this study the item 'My life as a whole' will be used, ratings ranges from 1= very dissatisfied to 6= very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Brogårdh, Principal Investigator — Department of Health Sciences, Faculty of Medicine, Lund University
Locations (1):
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carlsson H, Rosen B, Bjorkman A, Pessah-Rasmussen H, Brogardh C. SENSory re-learning of the UPPer limb (SENSUPP) after stroke: development and description of a novel intervention using the TIDieR checklist. Trials. 2021 Jul 5;22(1):430. doi: 10.1186/s13063-021-05375-6. PMID 34225764
- [Derived] Carlsson H, Rosen B, Pessah-Rasmussen H, Bjorkman A, Brogardh C. SENSory re-learning of the UPPer limb after stroke (SENSUPP): study protocol for a pilot randomized controlled trial. Trials. 2018 Apr 17;19(1):229. doi: 10.1186/s13063-018-2628-1. PMID 29665842